CLINICAL TRIAL: NCT03565718
Title: The Plant-Based and Soul-Full Study: Increasing African American Adults' Perceived Benefits of Consuming Plant-Based Foods
Brief Title: The Plant-Based and Soul-Full Study (PASS)
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00076585
Record Dates: First submitted 2018-06-04; First posted 2018-06-21 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Dietary Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): Participants in this group will receive counseling, informational materials, and recipes for following a vegan diet. Participants in this group will receive gift cards to go shopping at their local supermarkets and follow the diet for 3 weeks. At the end of the 3 week period each participant will have a follow-up meeting and provide feedback to the study personnel. The Dietary Intervention: Standard/Grocery includes intervention meetings and dietary counseling.
  Interventions: Behavioral: Dietary Intervention: Standard/Grocery
- Restaurant Group (Experimental): Participants in this group will receive counseling, informational materials, and recipes for following a vegan diet. Participants in this group will receive gift cards to go and eat out a few times a week at local vegan soul food restaurants and follow the diet for 3 weeks. At the end of the 3 week period each participant will have a follow-up meeting and provide feedback to the study personnel.
  The Dietary Intervention: Restaurant condition includes intervention meetings and dietary counseling.
  Interventions: Behavioral: Dietary Intervention: Restaurant

INTERVENTIONS:
Behavioral: Dietary Intervention: Restaurant — Participants will receive instruction on how to follow a vegan diet for three weeks and will receive gift cards to local vegan soul food restaurants.
  Arms: Restaurant Group
Behavioral: Dietary Intervention: Standard/Grocery — Participants will receive instruction on how to follow a vegan diet for three weeks and will receive gift cards to grocery stores.
  Arms: Standard Group

SUMMARY:
The goal of this study is to examine if exposure to vegan soul food restaurants can increase African American adults' perceived benefits of consuming plant-based foods more so than standard guidelines. Although the health benefits of vegan diets are well documented, many people are reluctant to commit to a vegan diet long term. Various issues like food preparation, a lack of social support, or other barriers are often mentioned as reasons why people can't be vegan. This study will (1) find out if short term exposure (i.e. 3 weeks) to culturally tailored curriculum focusing on the health benefits of consuming plant-based foods increases African American adults' perceptions of adopting a vegan diet. And (2) if eating out a few times a week at vegan soul food restaurants can further increase African American adults' perceived benefits of a vegan than having to prepare all meals at home.

DETAILED DESCRIPTION:
The goal of this study is to examine if exposure to vegan soul food restaurants can increase African American adults' perceived benefits of consuming plant-based foods more so than standard guidelines. Although the health benefits of vegan diets are well documented, many people are reluctant to commit to a vegan diet long term. Various issues like food preparation, a lack of social support, or other barriers are often mentioned as reasons why people can't be vegan. This study will (1) find out if short term exposure (i.e. 3 weeks) to culturally tailored curriculum focusing on the health benefits of consuming plant-based foods increases African American adults' perceptions of adopting a vegan diet. And (2) if eating out a few times a week at vegan soul food restaurants can further increase African American adults' perceived benefits of a vegan than having to prepare all meals at home.

Study participants will receive counseling and informational materials from a trained research assistant to follow a vegan diet for 3 weeks. Participants will be randomly assigned to either a standard group or a restaurant group. The standard group will receive gift cards to shop at local super markets. The restaurant group will receive gift cards to eat out a few times a week at local vegan soul food restaurants. Changes in individuals' perceived benefits and barriers to consuming plant-based foods will be assessed with a validated survey at baseline and at the end of the 3 week period.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Be between the ages of 18-65 years
* Live in the Columbia, SC/Midlands area
* Be able to attend all meetings with the study coordinator
* Be willing to be randomized to either condition

Exclusion Criteria:

* Currently following a vegan diet
* Under the age of 18 years old
* Over the age of 65 years old
* Not willing to attend meetings with the study coordinator
* Not willing to be randomized to either condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Dietary acceptability using the Food Acceptability Questionnaire | Baseline and three weeks
  Changes in acceptability of plant-based diets via a validated questionnaire

SECONDARY OUTCOMES:
Body weight using a digital scale | Baseline and three weeks
  Body weight assess objectively via calibrated digital scale.
Perceptions of Plant-based diets using the Perceived Barriers and Benefits Questionnaire | Baseline and three weeks
  Changes in perceptions of plant-based diets via a validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, Principal Investigator — University of Southern California
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided